CLINICAL TRIAL: NCT02293785
Title: GREAT (Good Response With Appropriate Treatment) "Factors Influencing the Analgesic Response Over Time of the Oxycodone-Naloxone Association in Painful Cancer Patients"
Brief Title: GREAT - Good Response With Appropriate Treatment
Status: Completed | Type: Observational
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Other Study IDs: DOL-IRFMN-6554
Record Dates: First submitted 2014-11-13; First posted 2014-11-18 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-03

CONDITIONS: Cancer Pain; Neoplasms
MeSH Terms: conditions — Cancer Pain; Neoplasms | interventions — oxycodone naloxone combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Oxycodone-Naloxone

SUMMARY:
The symptoms associated in advanced cancer patients and adverse events due to use of opioids have major influence on the state of health and quality of life of patients. The pain, in particular, is a symptom with severe negative impact and with a prevalence ranging between 33% and 64%, according to the stage of the disease, with values around 70-90% in advanced stages and metastatic.

The use of opioids, however, is usually associated with the appearance of common adverse events as drowsiness/sedation, constipation, nausea/vomiting, and dizziness. Some effects are self-limiting in the time for the appearance of tolerance while others, as constipation persist.

Several clinical studies have demonstrated that the association oxycodone-naloxone (OXN), which consists in the union between a molecule agonist and an antagonist of opioid receptors, reduced the constipation in the presence of unchanged analgesic efficacy compared to oxycodone alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnostic (histological or cytological) evidence of locally advanced or metastatic solid tumour;
* With average pain intensity > 4, measured with NRS and related to the last 24 hours, due to the cancer, requiring OXN for the first time;
* With life expectancy > one month;
* Strong opioid naïve;
* Eligible to take any of the medications under evaluation;
* With age ≥ 18 years.

Exclusion Criteria:

* With presence of other diseases, including psychiatric/mental illness, severe senile or other form of dementia, that can interfere with participation and compliance with the study protocol or can contraindicate the use of the investigational drugs;
* Diagnosis of primary brain tumor or leukaemia;
* Diagnosis of chronic renal failure;
* Patients with antalgic radiotherapy or radio-metabolic therapy in progress or completed less than 14 days before study;
* Patients starting a first line chemotherapy simultaneously to the beginning of the study;
* Other types of analgesic treatments, including local-regional anesthetic techniques or neurosurgical /ablative methods;
* Patients who cannot guarantee regular follow-up visits for logistic or geographic reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study involves a pain longitudinal evaluation in cancer patients through a follow-up of 4 weeks, which will examine in a dynamic clinical, biological and genetic aspects.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
non responders | 28 days
  Subjects will be classified as non-responders (NR) to treatment if between from the first and to last visit during the follow-up will not exhibit a reduction in average pain at least 30% and/or do not reach a final score of ≤ 4 pain points, defined as average pain experienced in the last 24 hours and measured by an 11-point numerical scale from 0 (no pain) to 10 (maximum pain imaginable).

SECONDARY OUTCOMES:
Opioids Escalation Index | 28 days
  Percentage of subjects that will need during the follow-up an increase in daily opioid dose ≥5%, measured by the OEI% (Opioids Escalation Index). The value of 5% identifies the cut-off between the increases of dose considered normal or high entity.
additional opioid treatment | 28 days
  Proportion of subjects that will need during the follow-up of an action to "additional" opioid treatment, in addition to the basic treatment programmed, to maintain the analgesic response in the treatment "around the clock".

CONTACTS AND LOCATIONS:
Locations (18):
- Italy (18):
  - Ospedale degli Infermi di Biella, Biella, Biella
  - IRCCS Centro di Riferimento Oncologico di Aviano, Aviano
  - Ospedale Oncologico A. Businco, Cagliari
  - E.O. Ospedali Galliera Genova, Genova
  - Presidio Ospedaliero di Macerata, Macerata
  - IRCCS Fondazione Cà Granda Ospedale Maggiore Policlinico di Milano, Milan
  - Istituto Scientifico San Raffaele, Milan
  - Ospedale di Mirano, Mirano
  - Ospedale V. Monaldi, Napoli
  - IRCCS Istituto Oncologico Veneto, Padua
  - Ospedale di Piacenza, Piacenza
  - Fondazione PTV Policlinico Tor Vergata, Roma
  - Ospedale San Camillo Forlanini, Roma
  - Policlinico Umberto I Università Sapienza, Roma
  - Policlinico Umberto I, Roma
  - A.O. Valtellina e Valchiavenna, Sondalo
  - Ospedale SS Trinità - Sora, Sora
  - Hospice "Raggio di Sole" SPA TP2, Trapani

REFERENCES:
- [Background] Corli O, Montanari M, Greco MT, Brunelli C, Kaasa S, Caraceni A, Apolone G. How to evaluate the effect of pain treatments in cancer patients: results from a longitudinal outcomes and endpoint Italian cohort study. Eur J Pain. 2013 Jul;17(6):858-66. doi: 10.1002/j.1532-2149.2012.00257.x. Epub 2012 Dec 5. PMID 23213042